CLINICAL TRIAL: NCT01861665
Title: A Comparative Trial of Marcaine Administration in Laparoscopic Gynecologic Surgery Using Either a Pre- or Post-operative Injection.
Brief Title: Marcaine Use in Laparoscopic Gynecological Surgery
Acronym: Marcaine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator no longer recruiting subjects.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 1004010977
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Post-operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients are acting as their own control receiving Bupivicaine (Marcaine) on both sides. One arm is pre incision the other arm is post incision.
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Marcaine administered pre-incision. (Active Comparator): Pre-operative administration, using both the specific drug - Marcaine 0.25%- and total amount - 5cc per incision.
  Interventions: Drug: Marcaine- 0.25%
- Marcaine administered post-incision (Active Comparator): Marcaine 0.25% administered post-incision, total amount 5cc per incision.
  Interventions: Drug: Marcaine 0.25%.

INTERVENTIONS:
Drug: Marcaine- 0.25% — Marcaine 0.25% administered pre-incision.
  Arms: Marcaine administered pre-incision.
Drug: Marcaine 0.25%. — Marcaine 0.25% administered post-incision.
  Arms: Marcaine administered post-incision

SUMMARY:
The purpose of this trial is to compare incisional pain in patients receiving pre-incisional versus post operative Marcaine injection.

DETAILED DESCRIPTION:
Post-operative pain control is a key component of a patient's experience with surgery. In laparoscopic surgery, small (5 to 12mm) incisions are made, usually at the umbilicus and/on at either side of the lower abdomen, to allow insertion of a laparoscopic camera ("scope") and various laparoscopic instruments. The advantages for the patient of this approach compared to conventional open surgery include faster recovery with a significantly shorter hospital stay, less pain and less requirements for pain medication with a better cosmetic outcome. In many cases, the patient will go home within 24 hours of surgery. Many laparoscopic surgeons administer local anesthesia at the incision sites to assist in post-operative pain control. The best method for administration of the local anesthetic for optimal pain relief remains unclear. Some research has demonstrated that perhaps preemptive administration of local anesthetic improves post-operative pain control although in these studies, differences in patient populations and perception of pain between different patients makes comparison difficult. Optimizing analgesia protocols would benefit patients resulting in better pain relief and less use of narcotic analgesics with their associated side effects.

ELIGIBILITY:
Inclusion Criteria:

* • Ages 18-50

  * BMI 20-35
  * Gynecologic ambulatory cases only
  * Total of 3 incisions, with left and right incisions both being 5mm-10mm in size
  * Not taking pain medications prior to surgery
  * Length of surgery up to 3 hours
  * PACU stay up to 6 hours
  * Willing and able to sign informed consent

Exclusion Criteria:

* • Age or BMI out of range

  * Surgery longer than 3 hours or PACU stay longer than 6 hours
  * patients with chronic pelvic pain
  * Oncologic cases
  * Pregnant patients

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Medical College of Cornell
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Result] Singer T, Huang JY, Schattman GL, Joseph M, Stubbs RE, Rosenwaks Z. RCT- Comparing Bupivicaine Adminstration in Laparoscopic Gynecologic Surgery Using Either a Pre-Incision or Post-Closure Injection. Journal of Minimally Invasive Gynecology 19 (6): S46, 2012.

RESULTS

PARTICIPANT FLOW:
Groups:
- Medication Pre Incision Left Med Post Incision Right: Subjects acted as their own control with the left side being injected with the medication pre incision and the right side being injected with medication post incision.
- Medication Pre Incision Right Med Post Incision Left: Subjects acted as their own control with right side being injected with the medication pre incision and left side being injected with the medication post incision.
Period: Overall Study
Arm/Group | Medication Pre Incision Left Med Post Incision Right | Medication Pre Incision Right Med Post Incision Left
Started | 10 | 17
Completed | 10 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Medication Pre Incision Left Med Post Incision Right: Participants acted as their own control with left side being injected with medication pre incision and right side being injected with medication post incision.
- Medication Pre Incision Right Med Post Incision Left: Participants acted as their own control with right side being injected with medication pre incision and left side being injected with medication post incision.
- Total: Total of all reporting groups
Arm/Group | Medication Pre Incision Left Med Post Incision Right | Medication Pre Incision Right Med Post Incision Left | Total
Number analyzed (Participants) | 10 | 17 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 17 | 27
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.6 (5.79) | 30.92 (3.87) | 32.26 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 17 | 27
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10 | 17 | 27

OUTCOME MEASURES:

1. Primary Outcome: Wong-Baker Faces Pain Rating Scale
Description: Pain level on post op day 1 and 2 study hypothesize will be less if Marcaine is administered pre instead of post incision. The pain scale is a numeric pain rating scale from 0-5, with zero being no pain and 5 being the worst pain imaginable, faces depicting no pain to worst pain.
Time Frame: Post surgery day 0, post surgery day 1, post surgery day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Marcaine Administered Post Incision: Post-operative administration, using both the specific drug - Marcaine 0.25%- and total amount - 5cc post incision.
  Marcaine- 0.25%: Marcaine 0.25% administered post-incision.
Arm/Group | Marcaine Administered Pre-incision | Marcaine Administered Post Incision
Number analyzed (Participants) | 27 | 27
units on a scale
  Post Op day 0 | 1.675 (1.39) | 1.6 (1.42)
  Post Op day 1 | 2 (0.97) | 1.85 (1.45)
  Post Op day 2 | 1 (1.6) | 0.75 (0.65)
Statistical Analysis 1: Comparison: Marcaine Administered Pre-incision vs Marcaine Administered Post Incision; Test type: Superiority; p = 0.8379, t-test, 2 sided — Pre Incision vs. Post Incision on Post op day 0
Statistical Analysis 2: Comparison: Marcaine Administered Pre-incision vs Marcaine Administered Post Incision; Test type: Superiority; p = 0.7263, t-test, 2 sided — Pre incision vs. Post incision post op day 1
Statistical Analysis 3: Comparison: Marcaine Administered Pre-incision vs Marcaine Administered Post Incision; Test type: Superiority; p = 0.5, t-test, 2 sided — Pre incision vs. Post incision day 2

ADVERSE EVENTS:
Time Frame: Adverse event data was monitored up to two weeks post op.
Arm/Group | Marcaine Administered Pre-incision. | Marcaine Administered Post-incision
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes